CLINICAL TRIAL: NCT07012408
Title: Muscle Injury Return To Play Design in Football; Effects of Backward Design Versus Forward Design . A Randomized Controlled Trial
Brief Title: Muscle Injury RTP Design in Football; Effects of Backward Design vs Forward Design.
Acronym: MIRTPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de les Illes Balears (Other)
Responsible Party: Principal Investigator, Oscar Vicente Rodriguez, Principal Investigator, Universitat de les Illes Balears
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UniversitatBalears
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Muscle Injuries; Football Players
Keywords: Return to play; Design; effects

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, single-center controlled clinical trial. There will be two groups: a control group and an intervention group.
  The study will be carried out in the work environment of the principal investigator and doctoral student at the University of the Balearic Islands (UIB) and Club Atlético de Madrid. The study will focus on the first and B teams, which are based at the Ciudad Deportiva del Cerro del Espino in Majadahonda, Madrid. The study will be included in the principal investigator's doctoral thesis.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): The intervention group: Subjects with muscle injuries who are assigned to this group will follow a return-to-play program with a progressive design.
  Interventions: Other: Return to play program with progressive design
- Control Group (Experimental): Control Group: The subjects (muscle injuries) that are assigned to this group will follow a Return to Play program with regressive design.
  Interventions: Other: Return to play program with regressive design

INTERVENTIONS:
Other: Return to play program with progressive design — This design has more open objectives than the regressive design. In the progressive design, the duration of the return-to-play program is not determined by a future date, but rather by the player's daily progress. This design is less commonly used for scheduling tasks and planning work. It is intended to be compared with the regressive design to determine which is more appropriate.
  Other Names: IG
  Arms: Intervention Group
Other: Return to play program with regressive design — Control Group: Subjects with muscle injuries assigned to this group will follow a Return to Play program with a regressive design. This design has fixed times and objectives from the beginning of the program to predict the athlete's exact discharge time. This design is commonly used for scheduling tasks and planning work. It is intended to evaluate the benefits and drawbacks of the design and compare them with those of the progressive design to determine which is more appropriate.
  Other Names: CG
  Arms: Control Group

SUMMARY:
Introduction

"Return-to-play" (RTP) is an English term that corresponds to "return to competition". It is important to understand that this return is a constant, dynamic, and personalized decision-making process . The main objective of RTP is not to predict the exact moment of an athlete's return; rather, it is to prevent new injuries. For this, adequate decision-making is necessary. There are several important steps in the process, including correct diagnosis, strict control of workloads, and intelligent management of modifiers intrinsic to the sport that can lead to anxiety and stress

How are the pieces of the RTP puzzle arranged and managed?

How are RTP processes evaluated today?

How should RTP be understood? Should it be understood statically, as a checklist, or as a constant decision-making process involving the player?

Main objective: Evaluate the design of the RTP process for muscle injuries in sports.

Specific objectives:

* To compare two RTP designs and evaluate how their design influences the anxiety experienced by the player.
* Identify variables that may be altered when choosing a regressive or progressive RTP design, such as sleep quality and cortisol level.
* To establish direction in the design of the RTP process.
* Create complete clinical guidelines on muscle injuries in sports with a focus on RTP design.

Material and Methods

Definition of the Study Subjects

The subjects of the study will be all players belonging to the first or B team who suffer a muscle injury diagnosed by magnetic resonance imaging. At the time of injury, they will be randomly assigned to either the control group (following a regressive RTP design) or the intervention group (following a progressive RTP design). Masking will be double-blind. The sample size will be N=74.

The secondary variables will be recorded in the database after diagnosis by MRI. Subsequently, the primary variables will be measured and recorded at the beginning, middle, and end of the RTP period.

It is estimated that approximately half of the necessary sample size has been reached: about 37 subjects with muscle injury. The first statistical analysis will then be carried out to observe the preliminary results.

After three years, once the analysis has been completed, the results and conclusions will be written up for publication in a journal.

DETAILED DESCRIPTION:
Capturing and Recruiting Participants

Since the players are from the same club and suffer muscle injuries, they will be included in the control and intervention groups for three years. The following section will explain that the sampling technique is consecutive and that participants can take part in the study several times, as long as they have a muscle injury diagnosed by resonance. Relapses of the same injury or injuries in the same or different muscle groups will also be included in the sample. The head of the club's medical service and collaborating researcher, Dr. José María Villalón Alonso, will recruit the participants. After the diagnostic test (MRI) is performed and the diagnosis and prognosis are established, the participants will be handed over to the recovery specialists, who will design the RTP. The specialists and the participants (players) will be blinded in the same way.

Allocation Procedure/Randomization

Subjects (muscle injuries) have the same probability (50%) of being allocated to the control or intervention group, regardless of previous allocations.

Justification of Sample Size

A type of consecutive sampling will be carried out based on the average probability that a soccer player will suffer a muscular injury. On average, each player will suffer 0.6 muscular injuries per season. In a team of 25 soccer players, this translates to an average of 15 muscular injuries per season. By contrasting this data with the club's database, we can verify the accuracy of this estimate. According to this statistical data, the population from which we will extract the sample will be the total number of muscle injuries suffered by the two teams of Club Atlético Madrid over three years:

0.6 (injuries) x 50 (players) x 3 years = 90 muscle injuries. Using the Grammo sample calculator with a relative error of 5% and a 95% confidence interval, we will calculate the necessary sample size for the sample to be representative, which will be N = 74.

Statistical Analysis Plan:

Phase 1: Use Levene's test to check if the variances of the control and intervention groups are equal.

Phase 2: Use a t-test to determine if there is a significant difference between the means of the control and intervention groups, and to establish whether the null hypothesis (H0) or the alternative hypothesis (HA) is true.

Phase 3: Perform a bivariate study of the relationship between anxiety (dependent variable) and estimated prognosis (independent variable) using Pearson's correlation coefficient.

Phase 4: Conduct a multivariate study through multiple regression between the dependent variable, sleep quality, and the independent variables, age, type of affected tissue, and cortisol level.

Phase 5: Perform a multivariate study through simple linear regression between the dependent variable, anxiety, and the independent variable, previous injuries in the same musculature.

Ethical and Legal Aspects:

Compliance with the standards of Good Clinical Practice, the Declaration of Helsinki, the Oviedo Convention, and the Personal Data Protection and Guarantee of Digital Rights Act (LO 3/2018, December 5, 2018), as well as the regulations for managing clinical histories.

The investigator undertakes to comply with the aforementioned rules throughout the development of the research protocol, as well as in the presentation to this ethics committee, for which the investigator must provide a certificate of Good Clinical Practice (GCP). The collaborating investigators also have this GCP certificate.

Informed Consent Form:

The patient information sheet and informed consent form are both attached in Annexes 1 and 2.

The confidentiality of information collected in the context of the study is guaranteed.

Data Controller: Óscar Vicente Rodríguez TLF: 699 874 059 Email: oscarvicente90@gmail.com

Purpose of data collection: Clinical and epidemiological research.

Maximum period of data retention: The data will be kept for four years (three years for the duration of the study and one extra year for future research).

Processing, communicating, and transferring the personal data of all participating subjects will comply with the provisions of Organic Law 3/2018 of December 5 on the protection of personal data and the guarantee of digital rights.

In accordance with the aforementioned legislation, you may exercise your rights of access, rectification, deletion, opposition, and limitation of data processing. You may also transfer your data to an authorized third party (portability). For these requests, please contact the principal investigator responsible for processing at oscarvicente90@gmail.com or C/Moreno Torroba 10, 1o B, CP. 28220 Majadahonda, Madrid.

The data will be computerized and incorporated into an automated personal data system that complies with all security measures for restricted access, as described in this document.

To guarantee the confidentiality of the obtained information:

Your data and the sample will be identified by a code, and only the study physician and their collaborators will be able to relate this data to you and your medical history. Therefore, your identity will not be disclosed to anyone except in case of medical emergency or legal or administrative requirement.

Only the essential data necessary for the study will be transmitted to third parties and other countries. In no case will the data contain information that can directly identify you, such as your name, initials, address, or social security number. If this transfer occurs, it will be for the aforementioned study purposes and will guarantee confidentiality with at least the level of protection guaranteed by the legislation in force in our country.

Access to your personal information will be restricted to the study physiotherapist, collaborators, health authorities, the Balearic Islands Research Ethics Committee, and authorized personnel when required to verify the study's data and procedures, always maintaining confidentiality in accordance with current legislation.

You may contact the Spanish Data Protection Agency with any claims related to the processing of your personal data.

The handling of biological samples will be in accordance with Law 14/2007 and Royal Decree 1716/2011.

Saliva samples to determine cortisol levels will be collected at the Ciudad Deportiva Atlético de Madrid clinic on three occasions: at the beginning of the RTP, after the magnetic resonance imaging diagnosis, halfway through the established prognosis, and the day before the RTP ends. The analysis will be performed at the same clinic, where, at the end of the cortisol measurement, the saliva will be discarded and only the recorded cortisol value will be kept.

Any risks associated with the procedure used to collect these samples are covered by the study insurance.

The sample will be coded and treated confidentially throughout this study. A code will be used to link the sample to you, and only the investigator and his staff will be able to decipher it to preserve your identity.

If additional data or samples are needed, your physical therapist will contact you to request your cooperation.

You will be informed of the reasons and asked again for your consent if necessary.

It will not receive any economic benefits from the donation of samples or the transfer of provided data, nor will it have any rights to possible commercial benefits from discoveries resulting from the research.

The samples will be analyzed in the Ciudad Deportiva Atlético de Madrid laboratory and stored for four years in case additional analyses related to the study's objectives are necessary. The person responsible for the samples will be the study promoter during this process.

At the end of the research period, your sample may be:

* Destroyed
* Anonymized (i.e., the link between the sample and you will be completely destroyed so that neither the researcher nor any other team member will be able to identify to whom your sample belongs again).
* Incorporated into a collection managed by researcher Óscar Vicente Rodríguez at the Ciudad Deportiva Atlético de Madrid so that it can continue to be used in the "Stress and Muscle Injury" study and line of research. ́

Samples are stored in the Ciudad Deportiva Atlético de Madrid biobank for use in other research projects, which may be unrelated to the initial study for which consent was given. The biobank may provide samples to authorized projects, including those abroad, with prior approval from the scientific and ethics committees. You may contact the biobank to obtain information on projects in which your samples were used.

Insurance Policy or Justification of Absence for Experimental Studies

Mr. Óscar Vicente Rodríguez is the principal investigator and has the following identification number: 35.572.548, and is a member with no. 1224, is registered in the Collective Policy of Professional Civil Responsibility, to which the Official College of Physiotherapists of the Balearic Islands adheres, with number 531000009 from A.M.A. (Agrupación Mutual Aseguradora - La Mutua de los Profesionales Sanitarios). Annex 3.

Commitment to publishing the results

The principal investigator is committed to publishing the results, regardless of their nature, since there is no conflict of interest. This trial will be part of the doctoral student's (principal investigator) thesis, which guarantees the publication of the results to improve the design of the RTP process.

Financial report and source of financing

The project has no private funding other than the 3,235.45 euros provided by PI Oscar Vicente Rodriguez for the cortisol ELISA measurement kits, Oura rings, and tablets used to record expenses. The MRI and radiological report expenses are free for the club due to the entity's nature, with no conflict of interest. The same applies to the team of statisticians who can analyze the results. They are part of the UIB and collaborate with doctoral theses. This essay is one such work. Regarding the CEIm of the Balearic Islands, this trial is exempt from fees (see the documentation), as it is part of the UIB's Doctoral School studies.

ELIGIBILITY:
Inclusion Criteria:

* Male soccer players.
* Diagnosed with a muscle injury via magnetic resonance imaging (MRI) during the three year study period.
* They will all belong to the same club.
* Age will be between 18 and 40 years old.

Exclusion Criteria:

* Patients (Muscle injuries) that do not cause players to miss training or competitions.
* Patients voluntarily decide not to participate in the study or abandon the RTP process due to transfers or other exceptional causes.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study will only include injuries to male soccer players.
Enrollment: 74 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-03 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | It will be measured at the beginning, middle, and end of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  Player Anxiety During the Return-to-Play Process. GAD-7 Anxiety scale.
  This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively,of "not at all," "several days," "more than half the days," and "nearly every day."
  GAD-7 total score for the seven items ranges from 0 to 21.
  0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Sleep quality | It will be measured at the beginning, middle, and end of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  The quality of the player's sleep during the Return to Play process. This is measured with the Oura Ring, which uses a validated scale to quantify sleep quality.
  Oura's Sleep Score.
  85-100: Optimal sleep quality. 70-84: Good sleep quality. 60-69: Fair sleep quality. 0-59: Areas for improvement are needed.
Stress (cortisol) | It will be measured at the beginning, middle, and end of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  Stress (cortisol) during the return-to-play process. We will measure it with the ELISA salivary kit to see how this hormone, which is directly related to the stress experienced by the athlete, varies.
  Cortisol levels are typically measured in micrograms per deciliter (mcg/dL) and fluctuate throughout the day, with the highest levels in the morning and the lowest at night. Normal ranges vary depending on the time of day and the testing method (blood, urine, or saliva), but generally, a healthy individual will have cortisol levels between 10-20 mcg/dL in the early morning (6-8 am) and 3-10 mcg/dL around 4 pm
Heart Rate Variability | It will be measured at the beginning, middle, and end of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  Player Heart Rate Variability During the Return-to-Play Process. Ouraring device.
  Interpreting HRV Scores:
  High HRV (e.g., 70 or higher):
  Associated with good health, a balanced autonomic nervous system, and better adaptability.
  Moderate HRV (e.g., 50-70):
  May indicate a need for improvement in areas like sleep, stress management, or nutrition.
  Low HRV (e.g., below 50):
  May indicate increased risk of health problems and a need for addressing underlying issues.

SECONDARY OUTCOMES:
Age | It will be measured and registered in the data base at the beginning of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  Age of player who suffered the muscle injury
History of previous muscle injuries in the same muscle. | It will be determined and registered in the data base at the beginning of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  History (Yes or No) of previous muscle injuries in the same muscle that suffers the injury that is included in the study.
Type of tissue involved in the muscle injury. | It will be determined and registered in the data base at the beginning of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  The type of tissue involved in the muscle injury is indicated by the radiological report and the BAMIC scale.
The estimated medical prognosis of the player's discharge. | It will be determined and registered in the data base at the beginning of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  The estimated medical prognosis of the player's discharge is reported in the radiology report and categorized using the BAMIC scale.
  The British Athletics Muscle Injury Classification proposes a new system, based on the available evidence, which should provide a sound diagnostic base for therapeutic decision-making and prognostication. Injuries are graded 0-4 based on MRI features, with Grades 1-4 including an additional suffix 'a', 'b' or 'c' if the injury is 'myofascial', 'musculo-tendinous' or 'intratendinous'.
Weight | It will be measured and registered in the data base at the beginning of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  Player weight in the moment of start Return to play
Height | It will be measured and registered in the data base at the beginning of the return-to-play process. This will be done for all subjects (muscle injuries) included in the study during the three years of the trial.
  Height of player

CONTACTS AND LOCATIONS:
Overall Officials: Olga Velasco, Phd Physio, Study Director — University of Balearic Islands
Locations (1):
- University of Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Yes
As part of a doctoral program's research plan, this essay's IPD will be shared with the thesis directors. The IPD is confidential and is only for this research.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be shared at the midpoint of the trial as part of the preliminary statistical analysis and at the end of the trial for the final statistical analysis and writing of the results and conclusions. The IPD will be coded using the patient code; therefore, there is no possibility of data exposure.
Access Criteria: The principal investigator, the student in the Ph.D. program, the two thesis supervisors from the University of the Balearic Islands, and the group of statisticians from the same university who are in charge of the statistical analysis will have access to the IPD.

REFERENCES:
- [Result] Orchard JW, Chaker Jomaa M, Orchard JJ, Rae K, Hoffman DT, Reddin T, Driscoll T. Fifteen-week window for recurrent muscle strains in football: a prospective cohort of 3600 muscle strains over 23 years in professional Australian rules football. Br J Sports Med. 2020 Sep;54(18):1103-1107. doi: 10.1136/bjsports-2019-100755. Epub 2020 Feb 5. PMID 32024646
- [Result] Dhillon H, Dhillon S, Dhillon MS. Current Concepts in Sports Injury Rehabilitation. Indian J Orthop. 2017 Sep-Oct;51(5):529-536. doi: 10.4103/ortho.IJOrtho_226_17. PMID 28966376
- [Result] Dattilo M, Antunes HKM, Galbes NMN, Monico-Neto M, DE Sa Souza H, Dos Santos Quaresma MVL, Lee KS, Ugrinowitsch C, Tufik S, DE Mello MT. Effects of Sleep Deprivation on Acute Skeletal Muscle Recovery after Exercise. Med Sci Sports Exerc. 2020 Feb;52(2):507-514. doi: 10.1249/MSS.0000000000002137. PMID 31469710
- [Result] Tabor J, La P, Kline G, Wang M, Bonfield S, Machan M, Wynne-Edwards K, Emery C, Debert C. Saliva Cortisol as a Biomarker of Injury in Youth Sport-Related Concussion. J Neurotrauma. 2023 Feb;40(3-4):296-308. doi: 10.1089/neu.2022.0190. Epub 2022 Sep 21. PMID 35906800
- [Result] Gomez-Espejo V, Olmedilla A, Abenza-Cano L, Garcia-Mas A, Ortega E. Psychological readiness to return to sports practice and risk of recurrence: Case studies. Front Psychol. 2022 Sep 23;13:905816. doi: 10.3389/fpsyg.2022.905816. eCollection 2022. PMID 36211933
- [Result] Orchard J, Best TM, Verrall GM. Return to play following muscle strains. Clin J Sport Med. 2005 Nov;15(6):436-41. doi: 10.1097/01.jsm.0000188206.54984.65. PMID 16278548
- [Result] Hoy MK, Stache S Jr, Roedl JB. Hamstring Injuries: A Paradigm for Return to Play. Semin Musculoskelet Radiol. 2024 Apr;28(2):119-129. doi: 10.1055/s-0043-1778027. Epub 2024 Mar 14. PMID 38484764
- [Result] Wong S, Ning A, Lee C, Feeley BT. Return to sport after muscle injury. Curr Rev Musculoskelet Med. 2015 Jun;8(2):168-75. doi: 10.1007/s12178-015-9262-2. PMID 25742905
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Result] Pollock N, James SL, Lee JC, Chakraverty R. British athletics muscle injury classification: a new grading system. Br J Sports Med. 2014 Sep;48(18):1347-51. doi: 10.1136/bjsports-2013-093302. Epub 2014 Jul 16. PMID 25031367
- [Result] Hagglund M, Walden M, Ekstrand J. Previous injury as a risk factor for injury in elite football: a prospective study over two consecutive seasons. Br J Sports Med. 2006 Sep;40(9):767-72. doi: 10.1136/bjsm.2006.026609. Epub 2006 Jul 19. PMID 16855067
- [Result] Papacosta E, Nassis GP. Saliva as a tool for monitoring steroid, peptide and immune markers in sport and exercise science. J Sci Med Sport. 2011 Sep;14(5):424-34. doi: 10.1016/j.jsams.2011.03.004. Epub 2011 Apr 7. PMID 21474377
- [Result] Svensson T, Madhawa K, Nt H, Chung UI, Svensson AK. Validity and reliability of the Oura Ring Generation 3 (Gen3) with Oura sleep staging algorithm 2.0 (OSSA 2.0) when compared to multi-night ambulatory polysomnography: A validation study of 96 participants and 421,045 epochs. Sleep Med. 2024 Mar;115:251-263. doi: 10.1016/j.sleep.2024.01.020. Epub 2024 Jan 26. PMID 38382312
- [Result] Palsson TS, Rubio-Peiroten A, Domenech-Garcia V. Sleep deprivation increases pain sensitivity following acute muscle soreness. Sleep Med. 2023 Sep;109:75-81. doi: 10.1016/j.sleep.2023.06.010. Epub 2023 Jun 24. PMID 37423022
- [Result] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Result] Vileikyte L. Stress and wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):49-55. doi: 10.1016/j.clindermatol.2006.09.005. PMID 17276201
- [Result] Salom J. Readaptación tas las lesiones deportivas, tratamiento multidisciplinar basado en la evidencia. Madrid: Ed. Panamericana; 2020. ISBN 9788491103967
- [Result] Chia L, Taylor D, Pappas E, Hegedus EJ, Michener LA. Beginning With the End in Mind: Implementing Backward Design to Improve Sports Injury Rehabilitation Practices. J Orthop Sports Phys Ther. 2022 Dec;52(12):770-776. doi: 10.2519/jospt.2022.11440. PMID 36453072
- [Result] Isern-Kebschull J, Pedret C, Mecho S, Pruna R, Alomar X, Yanguas X, Valle X, Kassarjian A, Martinez J, Tomas X, Rodas G. MRI findings prior to return to play as predictors of reinjury in professional athletes: a novel decision-making tool. Insights Imaging. 2022 Dec 27;13(1):203. doi: 10.1186/s13244-022-01341-1. PMID 36575363
- [Result] Delvaux F, Rochcongar P, Bruyere O, Bourlet G, Daniel C, Diverse P, Reginster JY, Croisier JL. Return-to-play criteria after hamstring injury: actual medicine practice in professional soccer teams. J Sports Sci Med. 2014 Sep 1;13(3):721-3. eCollection 2014 Sep. No abstract available. PMID 25177206
- [Result] Miller MD, Arciero RA, Cooper DE, Johnson DL, Best TM. Doc, when can he go back in the game? Instr Course Lect. 2009;58:437-43. PMID 19385553
- [Result] Creighton DW, Shrier I, Shultz R, Meeuwisse WH, Matheson GO. Return-to-play in sport: a decision-based model. Clin J Sport Med. 2010 Sep;20(5):379-85. doi: 10.1097/JSM.0b013e3181f3c0fe. PMID 20818198
- [Result] Matheson GO, Shultz R, Bido J, Mitten MJ, Meeuwisse WH, Shrier I. Return-to-play decisions: are they the team physician's responsibility? Clin J Sport Med. 2011 Jan;21(1):25-30. doi: 10.1097/JSM.0b013e3182095f92. PMID 21200167
- [Result] Lempainen L, Mecho S, Valle X, Mazzoni S, Villalon J, Freschi M, Stefanini L, Garcia-Romero-Perez A, Burova M, Pleshkov P, Pruna R, Pasta G, Kosola J. Management of anterior thigh injuries in soccer players: practical guide. BMC Sports Sci Med Rehabil. 2022 Mar 18;14(1):41. doi: 10.1186/s13102-022-00428-y. PMID 35303927
- [Result] Balius R, Pedret C. Lesiones musculares en el deporte. Barcelona: Ed. Panamericana; 2013. EAN: 9788498357035
- [Result] Ekstrand J, Hagglund M, Walden M. Epidemiology of muscle injuries in professional football (soccer). Am J Sports Med. 2011 Jun;39(6):1226-32. doi: 10.1177/0363546510395879. Epub 2011 Feb 18. PMID 21335353
- [Result] Kristenson K, Bjorneboe J, Walden M, Andersen TE, Ekstrand J, Hagglund M. Injuries in male professional football: A prospective comparison between individual and team-based exposure registration. Scand J Med Sci Sports. 2016 Oct;26(10):1225-32. doi: 10.1111/sms.12551. Epub 2015 Sep 17. PMID 26376838
- [Result] Rogers DL, Tanaka MJ, Cosgarea AJ, Ginsburg RD, Dreher GM. How Mental Health Affects Injury Risk and Outcomes in Athletes. Sports Health. 2024 Mar-Apr;16(2):222-229. doi: 10.1177/19417381231179678. Epub 2023 Jun 16. PMID 37326145
- [Result] Pruna, Ricard. "Return to play: ¿Hacia dónde vamos? Esto no es un juego de adivinanzas". Apunts: Medicina de l'esport, 2016, vol.VOL 51, núm. 191, p. 109-12
- [Result] Pedret Carles, Balius Ramon. Lesiones musculares en el deporte. Actualización de un artículo del Dr. Cabot, publicado en Apuntes de Medicina Deportiva en 1965. Apunts. Medicina de l'Esport.. 2015;50. 10.1016
- See also: Muscle injury guide Return to play management from Football Club Barcelona — https://static.capabiliaserver.com/frontend/clients/barca/wp/wp-content/uploads/2019/03/105e3b07-muscle-guide-general-principles-of-return-to-play-from-muscle-injury.pdf
- See also: Return to play following injuries in pro football: insights into the real-life practices,progression strategies and reintegration processes — https://sportperfsci.com/wp-content/uploads/2023/01/SPSR180_Buchheit.pdf
- See also: How to Deal with Anxiety Around Return to Play — https://moveunitedsport.org/truesport-how-to-deal-with-anxiety-around-return-to-play/
- See also: Mentally Preparing Athletes to Return to Play Following Injury — https://appliedsportpsych.org/resources/injury-rehabilitation/mentally-preparing-athletes-to-return-to-play-following-injury/
- See also: Cortisol and Stress recovery in handball team — https://dialnet.unirioja.es/servlet/articulo?codigo=6140420

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT07012408/Prot_SAP_ICF_000.pdf